CLINICAL TRIAL: NCT06432049
Title: Clinical and Radiographic Outcome of Endocrown Restoring First Permanent Molar in Children: Clinical Randomized Study
Brief Title: Endocrown Restoring First Permanent Molar in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Ahmed Ismail Taha, lecturer, Kafrelsheikh University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: MKSU/22-11-4
Record Dates: First submitted 2024-05-16; First posted 2024-05-29 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Comparing Different Types of Restorations for Restoring Endodontically Treated Permanent First Molar in Children
Keywords: Endocrown; CAD-CAM; Children; Ceramic; Molars

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PMC (Experimental): endodontically treated molar restored with Stainless steel crown
  Interventions: Other: restoration for endodontically treated molar
- EMX (Experimental): endodontically treated molar restored with endocrown fabricated from CAD-CAM lithium disillicate
  Interventions: Other: restoration for endodontically treated molar
- COP (Experimental): endodontically treated molar restored with endocrown fabricated from CAD-CAM composite
  Interventions: Other: restoration for endodontically treated molar

INTERVENTIONS:
Other: restoration for endodontically treated molar — prefabricated stainless steel crown or endocrown

SUMMARY:
Clinical and radiographic evaluation of endodontically treated first permanent molars in thirty children restored with three different restorations over 12 months

DETAILED DESCRIPTION:
This study comprised 30 children, with age range of (10-13) years old, with endodontically treated first permanent molars. Participants were classified into three groups according to type and material of the final restoration. All selected children were assigned to either PMC group (n=10) restored with performed metal crowns (Stainless-steel Molar Crowns) , EMX group (n=10) endocrown fabricated from CAD-CAM lithium disilicate glass ceramic , COP group (n=10) endocrown fabricated from CAD-CAM reinforced composite. After cementation, all children were evaluated over one year; at one week post-operative, 6 and 12 months for the following criteria: radiographic findings, plaque index, periodontal index, parent satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Patient age ranging from 10-13 years old with closed apex.
* Normal occlusion without any para-functional habits.
* Decayed lower first molar.
* Supra-gingival margin was required after preparation.
* Absence of root fractures or cracks.

Exclusion Criteria:

* Difficulty to apply rubber dam for proper endocrown bonding.
* Lack of patient cooperation for post-operative recall and follow up.
* Bad oral hygiene

Ages: 10 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2022-12-05 (Actual); Primary Completion 2023-11-09 (Actual); Study Completion 2024-05-13 (Actual)

PRIMARY OUTCOMES:
number of participants with pathological changes in radiographs | 6 months
  periodical radiograph was used to evaluate all 30 participants for recurrent caries or periapical pathologic findings
degree of parent satisfaction with different restorations | 6 month
  evaluation of the extent of parent satisfaction with different type of restorations using a special scale; Each reponse was scored as follows; (5) strongly agree, (4) agree (3) neutral, (2) disagree and (1) strongly disagree.
rate of plaque accumulation on different type of restorations | 6 months
  plaque index evaluate the plaque accumulation around different type of restorations. this index involves:
  * Plaque index 0: No plaque is in the area adjacent to the gingiva.
  * Plaque index 1: There is a plaque in the form of a thin film on the gingival margin.
  * Plaque index 2: There is a visible plaque in the gingival pocket and gingival margin.
  * Plaque index 3: There is a dense plaque in the gingival pocket and on the gingival margin.
effect of different restoration on surrounding gingiva | 6 months
  gingival index was used to evaluate the gingival health surrounding restorationsThis index involves a scale from 0 to 3 for the buccal, lingual, mesial and distal surfaces that is scored as follows: 0 indicates healthy gums; 1 indicates slight color changes, light edema and no presence of bleeding on probing; 2 indicates edema with slight redness and bleeding on probing; and 3 indicates severe edema, redness, the presence of ulceration and a tendency for spontaneous bleeding.

SECONDARY OUTCOMES:
number of participants with pathological changes in radiographs | 1 year
  periodical radiograph was used to evaluate all 30 participants for recurrent caries or periapical pathologic findings
degree of parent satisfaction with different restorations | 1 year
  using a special scale; Each reponse was scored as follows; (5) strongly agree, (4) agree (3) neutral, (2) disagree and (1) strongly disagree.
rate of plaque accumulation on different type of restorations | 1 year
  plaque index evaluate the plaque accumulation around different type of restorations. this index involves:
  * Plaque index 0: No plaque is in the area adjacent to the gingiva.
  * Plaque index 1: There is a plaque in the form of a thin film on the gingival margin.
  * Plaque index 2: There is a visible plaque in the gingival pocket and gingival margin.
  * Plaque index 3: There is a dense plaque in the gingival pocket and on the gingival margin.
effect of different restoration on surrounding gingiva | 1 year
  gingival index was used to evaluate the gingival health surrounding restorationsThis index involves a scale from 0 to 3 for the buccal, lingual, mesial and distal surfaces that is scored as follows: 0 indicates healthy gums; 1 indicates slight color changes, light edema and no presence of bleeding on probing; 2 indicates edema with slight redness and bleeding on probing; and 3 indicates severe edema, redness, the presence of ulceration and a tendency for spontaneous bleeding.

CONTACTS AND LOCATIONS:
Locations (1):
- Kafr El Shaikh University, Kafr ash Shaykh, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
all data will be shared after publishing.

REFERENCES:
- [Derived] Taha AI, Saad AE. Clinical and radiographic outcomes of endocrowns fabricated from two different CAD-CAM materials versus stainless steel crowns in restoring first permanent molars in children: a randomized clinical trial. BMC Oral Health. 2025 Jul 8;25(1):1127. doi: 10.1186/s12903-025-06507-z. PMID 40629344